CLINICAL TRIAL: NCT05728515
Title: Pilot Clinical Evaluation of a Small-molecule Carbonic Anhydrase IX Targeting PET Tracer in Clear Cell Renal Cell Carcinoma
Brief Title: A Small-molecule Carbonic Anhydrase IX Targeting PET Tracer in Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NYPILOT
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET scan (Experimental): Patients will receive an intravenous injection of 68Ga-NY104
  Interventions: Drug: 68Ga-NY104

INTERVENTIONS:
Drug: 68Ga-NY104 — Patients will undergo PET/CT scans after receiving an intravenous injection of 68Ga-NY104
  Other Names: no other intervention name

SUMMARY:
The goal of this pilot clinical trial is to see the potential application of a CAIX targeted PET. tracer in patients with clear cell renal cell carcinoma. The main question[s] it aims to answer are:

* The biodistribution of the PET tracer
* Whether RCC lesions can be identified by the PET tracer Participants will undergo 68Ga-NY104 PET/CT scan and images will be reviewed by nuclear medicine specialists.

DETAILED DESCRIPTION:
PET/CT imaging of three patients using 68Ga-NY104 for medical reasons will be performed. Patients received an intravenous injection of 68Ga-NY104. Images will be obtained at 0.5 h, 1 h, and 2 h after injection. A comparative 18F-FDG PET/CT scan will also be performed if necessary. The study will be carried out on a time-of-flight PET/CT scanner. SUVmax and SUVmean of normal organs and lesions, as well as tumor-to-background ratios, will be quantitatively assessed using a region-of-interest technique.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed or suspected metastatic ccRCC
2. Age ≥ 18 y
3. Written informed consent provided for participation in the trial
4. In the opinion of investigator, willing and able to comply with required study procedures.

Exclusion Criteria:

1. Patients on VEGF TKI treatment < 1 week before 68Ga-NY104 PET/CT. TKI is known to affect girentuximab binding in patients with ccRCC. If patients were on VEGF TKI treatment, such as sunitinib, sorafenib, cabozantinib, pazopanib, or lenvatinib, a washout of one week before 68Ga-NY104 PET/CT is required.
2. Pregnancy or breastfeeding.
3. Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 68Ga-NY104 in normal organs | From study completion to 2 hour after completion
  Uptake measured by SUVmax and SUVmean in normal organs using a region-of-interest technique
Tumor uptake of 68Ga-NY104 | From study completion to 2 hour after completion
  Uptake measured by SUVmax and SUVmean in suspected tumor lesions

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Images and quantitative measures will be available upon on request

REFERENCES:
- [Derived] Zhu W, Li X, Zheng G, Bai C, Ji Z, Zhang H, Xing H, Zhang Y, Huo L. Preclinical and pilot clinical evaluation of a small-molecule carbonic anhydrase IX targeting PET tracer in clear cell renal cell carcinoma. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):3116-3125. doi: 10.1007/s00259-023-06248-7. Epub 2023 May 29. PMID 37246998